CLINICAL TRIAL: NCT02776215
Title: Open-label Study to Investigate the Pharmacokinetics and Safety of Tasimelteon in Children and Adolescents
Brief Title: Study of the Pharmacokinetics and Safety of Tasimelteon in Children and Adolescents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VP-VEC-162-4201
Record Dates: First submitted 2016-05-16; First posted 2016-05-18 (Estimated); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Circadian Rhythm Sleep Disorders; Non-24 Hour Sleep-Wake Disorder; Autism Spectrum Disorder; Smith-Magenis Syndrome
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm; Autism Spectrum Disorder; Smith-Magenis Syndrome | interventions — tasimelteon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pharmacokinetic Dosing (Experimental): Single-dose pharmacokinetics of tasimelteon
  Interventions: Drug: tasimelteon

INTERVENTIONS:
Drug: tasimelteon — Melatonin receptor agonist
  Other Names: Hetlioz

SUMMARY:
Open-label Study to Investigate the Pharmacokinetics and Safety of Tasimelteon in Children and Adolescents.

DETAILED DESCRIPTION:
This study is an open-label, single dose, non-controlled study to evaluate the PK and safety of tasimelteon in children and adolescents from 3 years to less than 18 years of age who were legally blind and met the diagnostic criteria for CRSWD Non-24 per DSM-V or who were diagnosed with a Neurodevelopmental Disorder (like ASD and SMS) and had a nighttime sleep complaint.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females 3 to <18 years of age who are legally blind [defined as having a visual acuity of 20/200 or less in the better-seeing eye with best conventional correction (glasses or contact lenses) and/or a visual field of 20 degrees or less in the better-seeing eye], males or females 3 to <18 years of age with SMS and with a nighttime sleep complaint and males or females 3 to <18 years of age with ASD and with a nighttime sleep complaint;
2. Weigh at least 10 kg;

3 Diagnosis of SMS determined by a prior positive genetic test result as indicated by parent/guardian; Diagnosis of ASD as indicated by parent/guardian; or a diagnosis of Non-24 as determined by DSM-5 diagnostic criteria for the Circadian rhythm sleep-wake disorder, Non-24-hour sleep-wake hour type:

1. A persistent or recurrent pattern of sleep disruption that is primarily due to an alteration of the circadian system or to a misalignment between the endogenous circadian rhythm and the sleep-wake schedule required by an individual's physical environment or social or professional schedule;
2. The sleep disruption leads to excessive sleepiness or insomnia, or both;
3. The sleep disturbance causes clinically significant distress or impairment in social, occupational, and other important areas of functioning.

Exclusion Criteria:

1. For blind subjects only: Subjects who have a probable diagnosis of a current sleep disorder other than Non-24-Hour Sleep-Wake Disorder that is the primary cause of the sleep disturbance based on clinical investigator medical judgment;
2. For blind subjects only: History (within the 12 months prior to screening) of psychiatric disorders including ADHD, Neurodisabilities, Major Depressive Disorder, Generalized Anxiety Disorder, Axis II Disorders, delirium or any other psychiatric disorder, that is not being successfully treated or has not been resolved and that in the opinion of the clinical investigator would affect participation in the study or full compliance with study procedures;
3. History of intolerance and/or hypersensitivity to melatonin or melatonin agonists;

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2016-10-04 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Area under the curver (AUC) of tasimelteon and its metabolites | Pre-dose, 15 minutes post dose, 30 minutes post dose,1 hour post dose, 2 hours post dose, 4 hours post dose
Maximum concetration (Cmax) of tasimelteon and its metabolites | Pre-dose, 15 minutes post dose, 30 minutes post dose,1 hour post dose, 2 hours post dose, 4 hours post dose
Steady-state concentration (Css) of tasimelteon and its metabolites | Pre-dose, 15 minutes post dose, 30 minutes post dose,1 hour post dose, 2 hours post dose, 4 hours post dose
Half-life of tasimelteon and its metabolites | Pre-dose, 15 minutes post dose, 30 minutes post dose,1 hour post dose, 2 hours post dose, 4 hours post dose
Trough concentration (Ctrough) of tasimelteon and its metabolites | Pre-dose, 15 minutes post dose, 30 minutes post dose,1 hour post dose, 2 hours post dose, 4 hours post dose
Safety and tolerability of tasimelteon as measured by spontaneous reporting of adverse events (AEs) | Day 1
Safety and tolerability of tasimelteon as measured by Pediatric Adverse Event Reporting System (PAERS) | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Vanda Pharmaceuticals, Study Director — Sponsor GmbH
Locations (1):
- Parexel Early Phase Clinical Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No